CLINICAL TRIAL: NCT00740051
Title: A Randomised, db, Placebo-controlled, Parallel Group Efficacy and Safety Study of BI 1356 (5mg), Administered Orally Once Daily for 18 Weeks Followed by a 34 Week Double-blind Extension Period (Placebo Patients Switched to Glimepiride) in Type 2 Diabetic Patients With Insufficient Glycaemic Control for Whom Metformin Therapy is Inappropriate (Intolerability or Contraindication)
Brief Title: A Randomised, db, Placebo-controlled Study of BI 1356 for 18 Weeks Followed by a 34 Week Double-blind Extension Period (Placebo Patients Switched to Glimepiride) in Type 2 Diabetic Patients for Whom Treatment With Metformin is Inappropriate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.50; 2007-007485-38 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; glimepiride

ARMS (3):
- Linagliptin (Experimental): 52 week treatment
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): First 18 weeks of treatment
  Interventions: Drug: Linagliptin Placebo
- Glimepiride (Active Comparator): Placebo patients switch to glimepiride week19-52
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Linagliptin — 5mg once daily
  Arms: Linagliptin
Drug: Linagliptin Placebo — 0 mg placebo comparator for part 1 of study (to 18 weeks)
  Arms: Placebo
Drug: Glimepiride — 1-4mg for part 2 of study (weeks 19-52)
  Arms: Glimepiride

SUMMARY:
Efficacy of BI 1356 compared to placebo in patients for whom metformin therapy is inappropriate (intolerability, contraindication). The second part of the study looks at the safety of BI 1356 in this patient population with longer term treatment in comparison to a sulfonylurea drug (glimepiride)

ELIGIBILITY:
Inclusion criteria Patients between 18 and 80 years old with type 2 diabetes and insufficient glycemic control (HbA1c 7% to 10%) for whom metformin therapy is inappropriate (intolerability or contraindication)

Exclusion criteria Myocardial infarction, stroke or Transient ischaemic attack in last 6 months Treatment with rosiglitazone or pioglitazone, GLP-1 analogues, insulin or anti-obesity drugs in past 3 months Impaired hepatic function Severe renal impairment current treatment with systemic steroids change in dosage of thyroid hormones hereditary galactose intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (53):
- United States (15):
  - 1218.50.10009 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1218.50.10011 Boehringer Ingelheim Investigational Site, Peoria, Arizona
  - 1218.50.10013 Boehringer Ingelheim Investigational Site, Greenbrae, California
  - 1218.50.10016 Boehringer Ingelheim Investigational Site, Harbor City, California
  - 1218.50.10017 Boehringer Ingelheim Investigational Site, Huntington Park, California
  - 1218.50.10006 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.50.10007 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.50.10004 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1218.50.10002 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1218.50.10015 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1218.50.10005 Boehringer Ingelheim Investigational Site, Kingsport, Tennessee
  - 1218.50.10012 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.50.10022 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.50.10010 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.50.10018 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Canada (5):
  - 1218.50.11001 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1218.50.11003 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1218.50.11005 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.50.11002 Boehringer Ingelheim Investigational Site, Montague, Prince Edward Island
  - 1218.50.11004 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Mexico (9):
  - 1218.50.52007 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1218.50.52010 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1218.50.52009 Boehringer Ingelheim Investigational Site, León
  - 1218.50.52002 Boehringer Ingelheim Investigational Site, México
  - 1218.50.52004 Boehringer Ingelheim Investigational Site, México
  - 1218.50.52005 Boehringer Ingelheim Investigational Site, México
  - 1218.50.52008 Boehringer Ingelheim Investigational Site, México
  - 1218.50.52001 Boehringer Ingelheim Investigational Site, Monterrey
  - 1218.50.52003 Boehringer Ingelheim Investigational Site, Monterrey
- Philippines (9):
  - 1218.50.63003 Boehringer Ingelheim Investigational Site, Cebu
  - 1218.50.63005 Boehringer Ingelheim Investigational Site, Cebu
  - 1218.50.63006 Boehringer Ingelheim Investigational Site, Manila
  - 1218.50.63008 Boehringer Ingelheim Investigational Site, Manila
  - 1218.50.63001 Boehringer Ingelheim Investigational Site, Marikina City
  - 1218.50.63004 Boehringer Ingelheim Investigational Site, Marikina City
  - 1218.50.63007 Boehringer Ingelheim Investigational Site, Pasay
  - 1218.50.63002 Boehringer Ingelheim Investigational Site, Pasig
  - 1218.50.63009 Boehringer Ingelheim Investigational Site, Pasig
- Romania (5):
  - 1218.50.40004 Boehringer Ingelheim Investigational Site, Brasov
  - 1218.50.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1218.50.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1218.50.40005 Boehringer Ingelheim Investigational Site, Galati
  - 1218.50.40003 Boehringer Ingelheim Investigational Site, Sibiu
- Russia (5):
  - 1218.50.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.50.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.50.70002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.50.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.50.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Ukraine (5):
  - 1218.50.38002 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.50.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.50.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.50.38003 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.50.38005 Boehringer Ingelheim Investigational Site, Vinnitsa

REFERENCES:
- [Derived] Barnett AH, Patel S, Harper R, Toorawa R, Thiemann S, von Eynatten M, Woerle HJ. Linagliptin monotherapy in type 2 diabetes patients for whom metformin is inappropriate: an 18-week randomized, double-blind, placebo-controlled phase III trial with a 34-week active-controlled extension. Diabetes Obes Metab. 2012 Dec;14(12):1145-54. doi: 10.1111/dom.12011. Epub 2012 Oct 1. PMID 22974280
- [Derived] Johansen OE, Neubacher D, von Eynatten M, Patel S, Woerle HJ. Cardiovascular safety with linagliptin in patients with type 2 diabetes mellitus: a pre-specified, prospective, and adjudicated meta-analysis of a phase 3 programme. Cardiovasc Diabetol. 2012 Jan 10;11:3. doi: 10.1186/1475-2840-11-3. PMID 22234149
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/1218/1218.50_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Glimepiride: Patients treated with matching placebo (up to 18 weeks) followed by Glimepiride (after 18 weeks to 52 weeks)
- Linagliptin: Patients treated with Linagliptin 5mg once daily (up to 52 weeks)
Period: Overall Study
Arm/Group | Placebo/Glimepiride | Linagliptin
Started | 76 | 151
Completed | 58 | 119
Not Completed | 18 | 32
Not completed — Lack of Efficacy | 2 | 5
Not completed — Adverse Event | 1 | 4
Not completed — Protocol Violation | 2 | 6
Not completed — Lost to Follow-up | 3 | 8
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Other reason (not specified) | 4 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants and other baseline values taken from interim analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Glimepiride | Linagliptin | Total
Number analyzed (Participants) | 76 | 151 | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (9.7) | 56.4 (10.6) | 56.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 96 | 139
  Male | 33 | 55 | 88
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 30.19 (4.97) | 29.09 (5.62) | 29.46 (5.42)
Glycosylated hemoglobin (HbA1c) - Interim Analysis [Mean (Standard Deviation); unit: percent] — Baseline HbA1c was determined for the Full Analysis Set with a total of 73 patients treated with Placebo and 147 patients treated with Linagliptin (220 in total).
  percent | 8.06 (0.89) | 8.11 (0.95) | 8.09 (0.93)
Fasting blood plasma (FPG) glucose [Mean (Standard Deviation); unit: mg/dL] — Baseline fasting blood plasma glucose was determined for the Full Analysis Set with a total of 73 patients treated with Placebo and 147 patients treated with Linagliptin (220 in total).
  mg/dL | 180.5 (44.7) | 183.3 (46.4) | 182.4 (45.8)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 18 (Interim Analysis)
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the Week 0 HbA1c percent. Means are adjusted for baseline HbA1c, prior OADs and reason for metformin intolerance.
Time Frame: Baseline and week 18
Population: The Full Analysis Set (FAS) included all treated patients with a baseline and at least one on-treatment HbA1c measurement available during the first phase of the study. Last Observation Carried Forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: percent
Groups:
- Placebo: Patients treated with matching placebo (up to 18 weeks) followed by Glimepiride (after 18 weeks to 52 weeks)
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 73 | 147
percent | 0.14 (0.16) | -0.44 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin versus Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of p-values; Mean Difference (Final Values) = -0.57, 95% CI [-0.86 to -0.29], Standard Error of Mean 0.14

2. Primary Outcome: HbA1c Change From Baseline at Week 18 (Final Analysis)
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the Week 0 HbA1c percent. Means are adjusted for baseline HbA1c, prior OADs and reason for metformin intolerance. HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the Week 0 HbA1c percent. Means are adjusted for baseline HbA1c, prior OADs and reason for metformin intolerance. The primary analysis was re-run at the completion of the study in the final study report.
Time Frame: Baseline and week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 73 | 147
percent | 0.21 (0.16) | -0.39 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin versus Placebo. The primary analysis performed at the interim was re-run at the end of the study to accommodate changes made to the final study database; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of p-values; Mean Difference (Final Values) = -0.60, 95% CI [-0.88 to -0.32], Standard Error of Mean 0.14

3. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline at Week 18 (Interim Analysis)
Description: This change from baseline reflects the Week 18 FPG minus the Week 0 FPG. Means are adjusted for baseline FPG, baseline HbA1c, prior OADs and reason for metformin intolerance (Interim Analysis).
Time Frame: Baseline and week 18
Population: All patients in FAS with values for FPG at baseline and at week 18. Last Observation Carried Forward (LOCF) was used as the imputation rule (Interim Analysis).
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 66 | 138
mg/dl | 7.2 (6.0) | -13.3 (5.2)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin versus Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA — No adjustment of p-values; Mean Difference (Final Values) = -20.5, 95% CI [-31.1 to -9.9], Standard Error of Mean 5.4

4. Secondary Outcome: Percentage of Patients With HbA1c<7.0 at Week 18 (Interim Analysis)
Description: Odds ratios are adjusted for baseline HbA1c, prior OADs and reason for metformin intolerance.
Time Frame: Week 18
Population: Full Analysis Set (FAS) patients with baseline HbA1c >= 7.0%. Patients without a value at week 18 were analysed as non-responders.
Measure: Number; unit: percent of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 68 | 136
percent of patients | 11.8 | 23.5
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin versus Placebo; Test type: Superiority or Other; p = 0.0374, Regression, Logistic — No adjustment of p-values; Odds Ratio (OR) = 2.576, 95% CI [1.057 to 6.279]

5. Secondary Outcome: Percentage of Patients With HbA1c<6.5 at Week 18 (Interim Analysis)
Description: Odds ratios are adjusted for baseline HbA1c, prior OADs and reason for metformin intolerance.
Time Frame: Week 18
Population: FAS patients with baseline HbA1c >= 6.5%. Patients without a value at Week 18 were analysed as non-responders.
Measure: Number; unit: percent of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 70 | 146
percent of patients | 2.9 | 8.9
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p = 0.1281, Regression, Logistic — No adjustment of p-values; Odds Ratio (OR) = 3.285, 95% CI [0.710 to 15.196]

6. Secondary Outcome: Percentage of Patients With HbA1c Lowering by 0.5% at Week 18 (Interim Analysis)
Description: Odds ratios are adjusted for baseline HbA1c, prior OADs and reason for metformin intolerance.
Time Frame: Week 18
Population: The Full Analysis Set (FAS) included all treated patients with a baseline and at least one on-treatment HbA1c measurement available during the first phase of the study. Patients without a value at week 18 were analysed as non-responders.
Measure: Number; unit: percent of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 73 | 147
percent of patients | 17.8 | 36.1
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin versus Placebo; Test type: Superiority or Other; p = 0.0046, Regression, Logistic — No adjustment of p-values; Odds Ratio (OR) = 2.801, 95% CI [1.374 to 5.711]

7. Secondary Outcome: The Change in HbA1c From Baseline by Visit Over Time
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the HbA1c percent (at weeks 6, 12, 18, 22, 26, 30, 34, 40, 46, 52) minus the Week 0 HbA1c percent.
Time Frame: Baseline and weeks 6,12, 18, 22, 26, 30, 34, 40, 46, 52
Population: Treated set (OC)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo/Glimepiride | Linagliptin
Number analyzed (Participants) | 76 | 151
percent
  Change from baseline at week 6 (N=64, 136) | 0.26 (0.98) | -0.21 (0.77)
  Change from baseline at week 12 (N=57, 129) | 0.26 (1.08) | -0.43 (0.84)
  Change from baseline at week 18 (N=47, 118) | 0.10 (1.06) | -0.38 (0.87)
  Change from baseline at week 22 (N=46, 113) | -0.32 (0.82) | -0.40 (0.94)
  Change from baseline at week 26 (N=50, 110) | -0.53 (0.93) | -0.48 (0.92)
  Change from baseline at week 30 (N=49, 98) | -0.79 (1.06) | -0.49 (0.92)
  Change from baseline at week 34 (N=50, 96) | -0.75 (0.95) | -0.49 (0.88)
  Change from baseline at week 40 (N=49, 94) | -0.73 (1.11) | -0.45 (0.90)
  Change from baseline at week 46 (N=45, 92) | -0.78 (1.04) | -0.42 (0.96)
  Change from baseline at week 52 (N=45, 92) | -0.72 (1.01) | -0.44 (1.00)

8. Secondary Outcome: The Change in FPG From Baseline by Visit Over Time
Description: This change from baseline reflects the FPG (at weeks 6, 12, 18, 22, 26, 30, 34, 40, 46, 52) minus the Week 0 FPG.
Time Frame: Baseline and weeks 6,12,18, 22, 26, 30, 34, 40, 46, 52
Population: Treated set (OC)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo/Glimepiride | Linagliptin
Number analyzed (Participants) | 76 | 151
mg/dL
  Change from baseline at week 6 (N=63, 134) | 9.7 (30.7) | -8.4 (41.0)
  Change from baseline at week 12 (N=55,92) | 5.4 (33.0) | -14.3 (37.3)
  Change from baseline at week 18 (N=47, 115) | 5.0 (32.4) | -12.9 (35.9)
  Change from baseline at week 22 (N=46, 110) | -19.3 (33.3) | -14.0 (41.8)
  Change from baseline at week 26 (N=50, 108) | -22.6 (33.8) | -17.0 (37.8)
  Change from baseline at week 30 (N=48, 95) | -31.4 (29.5) | -19.1 (39.1)
  Change from baseline at week 34 (N=48, 95) | -25.6 (35.2) | -15.8 (36.0)
  Change from baseline at week 40 (N=47, 92) | -19.5 (33.2) | -19.0 (36.9)
  Change from baseline at week 46 (N=47, 92) | -22.8 (32.3) | -18.1 (38.8)
  Change from baseline at week 52 (N=43, 86) | -19.1 (30.1) | -14.0 (37.1)

ADVERSE EVENTS:
Time Frame: 52 weeks + 7 days
Description: These are the total results after the final completion of the study after 52 weeks. The time frame 52 weeks + 7 days (post-trt) is the maximum time frame. Some patients were not followed up for this long, and will correspondingly have had less opportunity to report the events.
Arm/Group | Placebo/Glimepiride | Linagliptin
Serious Adverse Events (participants affected / at risk) | 3/76 | 1/151
Other Adverse Events (participants affected / at risk) | 40/76 | 59/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Glimepiride (N=76) | Linagliptin (N=151)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Glimepiride (N=76) | Linagliptin (N=151)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 5 | 2
Influenza (Infections and infestations) | 2 | 8
Nasopharyngitis (Infections and infestations) | 6 | 15
Upper respiratory tract infection (Infections and infestations) | 7 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 22
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Dizziness (Nervous system disorders) | 4 | 11
Headache (Nervous system disorders) | 6 | 8
Anxiety (Psychiatric disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
Primary analysis (at interim) was rerun using final study database

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.